CLINICAL TRIAL: NCT06300333
Title: Effectiveness and Safety of a New Methotrexate Regimen in Treatment of Undisturbed Tubal Ectopic Pregnancy : A Pilot Prospective Study
Brief Title: Treatment of Ectopic Pregnancy by Low Dose of Methotrexate
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Mohamed Abouelhassan, principal invistigator, Assiut University
Other Study IDs: Ectopic tubal pregnancy
Record Dates: First submitted 2024-01-24; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Methotrexate — use low dose of Methotrexate in treatment of un distectopic tubal pregnancy

SUMMARY:
Evaluate the efficacy and safety of the use of low dose regimen of methotrexate in treatment of tubal undisturbed tubal ectopic pregnancy

DETAILED DESCRIPTION:
Ectopic pregnancy, also known as extrauterine pregnancy, occurs when the blastocyst implants outside the body of the uterus . The incidence is approximately 1.5-2.0 % of all pregnancies. The most frequent location for ectopic pregnancy is the uterine tube (96-98 %), followed by the cervix (0.2-0.5 %), the ovary (0.2-2.0 %), and the abdomen (˂1 %) . High-resolution ultrasonography and quantitative assessment of human chorionic gonadotropin (hCG) allow early diagnosis. Mortalities are now therefore rare, at 0.05 % of cases . Tubal pregnancy is the most frequent form and subject of the present article. Due to growth of the blastocyst, usually in the sixth to ninth gestational weeks, increasing wall tension develops in the uterine tube, with unilateral lower abdominal pain. If the uterine tube ruptures, intraabdominal bleeding may occur, with hematoperitoneum and possible hemorrhagic shock . The classic triad of symptoms-absence of menstruation, vaginal spotting, and lower abdominal pain-is often observed, but is not inevitable. The clinical findings can be extremely variable, ranging from symptom-free courses to the full picture of acute abdomen . Surgical treatment of tubal pregnancy is necessary in hemodynamically unstable patients and patients with acute pain or ultrasound evidence of free fluid in the abdomen. The standard surgical procedure is laparoscopic salpingotomy or salpingectomy . . Laparotomy is now only required in 1-2 % of patients with ectopic pregnancy. Tubepreserving surgery should always be aimed for, particularly in younger patients who are still planning to have children. Another treatment option is administration of methotrexate (MTX), a folic acid antagonist that blocks DNA/ RNA synthesis and thus cell division. In the single-dose protocol, methotrexate 50 mg/m2 body surface is administered on day 1 intramuscularly or intravenously , The hCG value is measured on days 4 and 7. If a drop in the hCG value by at least 15 % has not yet occurred, a second MTX dosage of 50 mg/m2 body surface should be administered. If there is a drop of[15 %, weekly hCG check-ups are carried out until the value is below the detection threshold of the relevant assay , Patients treated with the single dose require a second MTX injection in 13.5 % of cases, and less than 1 % required three or more MTX injections . However, there have been no dose-finding studies on the administration of MTX in patients with ectopic pregnancy, and several groups have reported good success rates of between 85.4 and 98.7 % using much lower dosages .the aim of this study is to use a low dose of Methotrexate in the treatment of tubal undisturbed ectopic pregnancy to get get less side e

ELIGIBILITY:
Inclusion Criteria:

* undisturbed ectopic tubal pregnancy Bhcg < 5000
* Haemodynamicaly stable
* Normal liver and kidney functions
* Commitment for fullow up untill ectopic pregnancy resolvede

Exclusion Criteria:

* disturbed ectopic pregnancy
* Bhcg >5000
* Persistent abdominal pain
* Lactating women
* women with abnormal liver and kidney functions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: the study will include women with undisturbed ectopic tubal pregnancy Bhcg < 5000 Haemodynamicaly stable Normal liver and kidney functions Commitment for fullow up untill ectopic pregnancy resolved
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
descriptive measurements of the results of using low dose methotrexate regimen in treatment of tubal undisturbed ectopic pregnancy | 7 day
  we will follow up cases by investigationssand ultrasound and describe the results of using the low dose methotrexate in treatment of tubal undisturbed ectopic pregnancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marion LL, Meeks GR. Ectopic pregnancy: History, incidence, epidemiology, and risk factors. Clin Obstet Gynecol. 2012 Jun;55(2):376-86. doi: 10.1097/GRF.0b013e3182516d7b. PMID 22510618
- [Background] Practice Committee of American Society for Reproductive Medicine. Medical treatment of ectopic pregnancy. Fertil Steril. 2008 Nov;90(5 Suppl):S206-12. doi: 10.1016/j.fertnstert.2008.08.049. PMID 19007632
- [Background] Karol D, Williamson M, Pereira N. Successful Expectant Management of a Tubal Ectopic Pregnancy. J Minim Invasive Gynecol. 2024 Feb;31(2):92-94. doi: 10.1016/j.jmig.2023.11.011. Epub 2023 Nov 30. No abstract available. PMID 38042476